CLINICAL TRIAL: NCT06257550
Title: THRIVE: AdapTive Personalized Dietitian coacHing, Messaging and pRoduce prescrIption to improVE Healthy Dietary Behaviors
Brief Title: AdapTive Personalized Dietitian coacHing, Messaging and pRoduce prescrIption to improVE Healthy Dietary Behaviors
Acronym: THRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00427492; 24FIM1264121 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2024-02-05; First posted 2024-02-14 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors and data analysts will be masked to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THRIVE Intervention Arm (Experimental): The THRIVE intervention arm will receive produce prescription, personalized dietitian coaching, adaptive bi-directional messaging; and linkages to social services.
  Interventions: Behavioral: THRIVE Intervention
- Comparator Arm (Active Comparator): The comparator arm will receive standard produce bags; and linkages to social services.
  Interventions: Behavioral: Active Comparator

INTERVENTIONS:
Behavioral: THRIVE Intervention — THRIVE Intervention includes:
  1. Weekly Pulse Surveys
  2. Adaptive culturally tailored messages
  3. Personalized Dietitian Coaching
  4. Produce Prescription "FARMacy" Mobile Market
  5. Linkages to Social Services
  Arms: THRIVE Intervention Arm
Behavioral: Active Comparator — The Active Comparator arm will receive standard produce bags through our food is medicine partner, and will receive the linkages to needed social and health resources intervention components.
  Arms: Comparator Arm

SUMMARY:
THRIVE intervention is a 2-arm randomized pilot trial testing the feasibility and preliminary efficacy of producing prescriptions, tailored dietitian counseling with adaptive messages, and linkages to social resources among 80 Black adults with hypertension.

DETAILED DESCRIPTION:
Nearly 55% of Black adults have hypertension and uncontrolled blood pressure. Dietary Approaches to Stop Hypertension (DASH) promotes a dietary pattern rich in fruits and vegetables (fruits and vegetables), low-fat dairy, lean meats with reduced saturated fat, and sweets, which is effective in lowering blood pressure. The proposed THRIVE intervention will enroll 80 Black adults with hypertension living in Healthy Food Priority Areas (HFPAs) in a 2-arm randomized pilot study. One group will receive Produce prescriptions, personalized dietitian coaching, and adaptive bi-directional messaging; the other group will receive standard produce bags. Both groups will be linked to needed social services.

The investigators will assess changes in overall DASH adherence, acceptability, and feasibility at 3- and 6-months post-randomization. The investigators will: 1) Develop and beta test THRIVE among Black adults with hypertension living in HFPAs; 2) Test feasibility and preliminary efficacy of THRIVE at 6 & 12 weeks; 3) Determine short-term sustainability of THRIVE at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Self-identify as Black/African American
3. Have diagnosed hypertension stages 1 (130-139/80-89 mm Hg) OR 2 (>140/90 mm Hg), determined via self-report and/or Electronic Medical Records (EMR)
4. Live in census tracts identified by Montgomery County Department of Planning as HFPA:

   1. Healthy Food Availability Index score is low (0-9.5),
   2. Median household income ≤185% of Federal Poverty Level
   3. >30% households have no vehicle, Distance to supermarket >1/4 mile.
5. Participants must have refrigeration, food appliances (microwave, stove),
6. Cell phone to receive messages

Exclusion Criteria:

1. Age <18 years
2. Type 1 or Type 2 Diabetes defined as a hemoglobin A1c ≥6.5% or diabetes treatment
3. Diagnosis of end-stage renal disease (ESRD)
4. Condition which interferes with outcome measurement (e.g., dialysis)
5. Serious medical condition which either limits life expectancy or requires active management (e.g. cancer)
6. Significant food allergies, preferences, intolerances, or dietary requirements that would interfere with diet adherence
7. Patients with cognitive impairment or other condition preventing their participation in the intervention
8. Current participation in a care management program related to health conditions (e.g., weight reduction, smoking cessation)
9. Current participation in another clinical trial that could interfere with the study protocol
10. Those planning to move out of the geographic area in 12 months
11. Unwillingness to provide informed consent
12. Other conditions or situations at the discretion of the Investigative team

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
DASH Adherence as assessed by the Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24) | 0, 12 weeks and 24 weeks
  Adherence will be assessed by the Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24). The scores range from 0 to 100, with higher scores reflecting greater adherence.

SECONDARY OUTCOMES:
Recruitment rate | 0, 12 weeks, 24 weeks
  Recruitment yield per time
Cost of the intervention | 0, 12 weeks, 24 weeks
  Intervention cost/person will be estimated based on the cost of the intervention
Participant Accrual | 0, 12 weeks and 24 weeks
  Referrals, participation rates, and recruitment yields.
Number of referrals to health and social need resources | 0, 12 weeks and 24 weeks
  Social needs as assessed by the number of participants connected to health services and services for social needs.
Systolic Blood pressure | 0, 12 and 24 weeks
  Blood pressure measured in millimeters of mercury (mmHg)
Diastolic Blood pressure | 0, 12 and 24 weeks
  Blood pressure measured in millimeters of mercury (mmHg)
Hemoglobin A1c | 0, 12 and 24 weeks
  Hemoglobin A1c (percent)
Height in inches | 0, 12 and 24 weeks
  Height will be measured
Weight in pounds | 0, 12 weeks and 24 weeks
  Weight will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Oluwabunmi Ogungbe, PhD, MPH, RN, Principal Investigator — JHU School Of Nursing
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States